CLINICAL TRIAL: NCT00377247
Title: Active Immunization of Patients With Carcinoma of Oral Cavity or Oropharynx With Autologous Dendritic Cells Transfected With DNA From Autologous Tumor (Phase I/II Study)
Brief Title: Active Immunization of Patients With Carcinoma of Oral Cavity or Oropharynx With Autologous Dendritic Cells Transfected With DNA From Autologous Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study closed to accrual due to slow accrual
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jonas Johnson, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-178; NIH R01-DE13818
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Primary Advanced Carcinoma of the Oral Cavity or Oropharynx; Squamous Cell Carcinoma of the Head and Neck
Keywords: Carcinoma; Head; Neck; Oral Cavity; Oropharynx; Mouth
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Cells w/Tumor DNA (Experimental)
  Interventions: Biological: autologous monocyte-derived dendritic cells (DC) transfected with DNA

INTERVENTIONS:
Biological: autologous monocyte-derived dendritic cells (DC) transfected with DNA — The patients will receive 1 x 107 DC/vaccine delivered intranodally or perinodally to lymph nodes (LN) distant from the head and neck area (e.g., to inguinal LN)

SUMMARY:
The primary goal of this study is to determine if the vaccine can be safely given to subjects, and to see what side effects occur (both good and bad) when they are given this experimental tumor vaccine. During this study, investigators intend to watch for tumor response while examining the effects of this vaccine on the body's immune system after it is given.

DETAILED DESCRIPTION:
This is an uncontrolled, non-randomized trial to evaluate safety, immunogenicity and feasibility of a new vaccine, consisting of autologous monocyte-derived dendritic cells (DC) transfected with autologous tumor-derived DNA. Briefly, the plan is to use a two-stage trial design and to initially enroll 17 patients with primary advanced carcinoma of the oral cavity or oropharynx over a period of 2 years. The patients will undergo surgery, and a portion of the primary tumor specimen not necessary for the pathologic diagnosis will be obtained to serve as a source of tumor DNA. Each DC-based vaccine will contain DNA-transfected DC. It will be administered intranodally under ultrasound guidance. Only those patients who have normal delayed type hypersensitivity (DTH) responses to recall antigens will be eligible to receive the vaccine. Immunologic response to the vaccine will be evaluated. If there is no evidence of toxicity, and >3 patients show immunologic response, the second stage of the study will be opened for accrual of 22 patients. All patients will be monitored by interferon- gamma (IFN-) secretion in enzyme-linked immunospot (ELISPOT) assays prior to and after vaccination for the frequency of T-cells responsive to autologous tumor and to the vaccine. The patients will also be evaluated before and after vaccination for the capability of their T cells to respond to activating signals delivered via the T cell receptor (TcR).

Primary Objective: To determine the safety and feasibility of immunization of patients with carcinoma of the oral cavity or oropharynx with autologous monocyte-derived dendritic cells (DC) transfected with DNA obtained from the patient's own cancer cells.

Secondary Objective: To evaluate the ability of the DNA-based DC vaccine to induce immune responses to the vaccine as well as to autologous tumor.

ELIGIBILITY:
Inclusion Criteria:

-

Written informed consent conforming to the institutional guidelines obtained from the patient.

Documented evidence of oral carcinoma or carcinoma of the oropharynx. Patients will undergo surgery, surgery and radiation or chemoradiation therapy, and will become eligible for the first vaccine between 1and 4 months after termination of conventional therapy.

Adequate immune competence, as indicated by positive reaction to one or more of the DTH skin tests.

Age 18 or above. Karnofsky performance status > 70% and life expectancy > eight months.

Adequate hematologic function:

Absolute neutrophil count > 1,000/mm3 Absolute lymphocyte count > 1,000/mm3 Hemoglobin > 9 g/dl Platelets > 100,000/mm3 h) Liver function tests: Bilirubin (total) < 1.7 mg/dl Alkaline phosphatase < 78 u/L (2 x ULN) SGOT < 54 u/L (2 x ULN) Lactic dehydrogenase < 180 u/L (2 x ULN) i) Kidney profile: Serum electrolytes Sodium 135-145 mEq/L Potassium 3.5-5.0 mEq/L Bicarbonate 21-28 mEq/L Chloride 100-108 mmol/L 2) Serum creatinine <4.5 mg/dL (3 x ULN) 3) BUN 8-25 mg/dL j) At least four weeks since any prior radiation therapy, immunotherapy, or chemotherapy

Exclusion Criteria:

- One or more of the Inclusion Criteria are not met. A significant history or current evidence of cardiac disease including, but not limited to, congestive heart failure, coronary artery disease, angina pectoris, uncontrolled hypertension, serious arrhythmias; or myocardial infarction within the previous six months.

Evidence of active infection requiring antibiotic therapy. Positive HIV or Hepatitis B or C screen tests Active intracranial metastases. Previously resected intracranial disease and or previously irradiated intracranial metastases which have been stable for four weeks are eligible.

History of other concurrent malignancies except basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.

Pregnant or lactating women. Patients requiring systemic corticosteroids (unless patient has had NO STEROIDS IN THE PAST 4 WEEKS).

Autoimmune disease including, but not limited to, rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, or ankylosing spondylitis

Min Age: 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety and feasibility of immunization of patients with the carcinomas of the oral cavity or the oropharynx with autologous DCs nucleofected with tumor DNA obtained from the patient's own tumor. | 6 months

SECONDARY OUTCOMES:
To determine whether the immunological responses to the vaccine and/or antitumor immune responses can be induced in patients who receive the vaccine | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonas T Johnson, M.D., Principal Investigator — UMPC/UPCI
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States